CLINICAL TRIAL: NCT01700361
Title: Visual Erotica, EMG, and Sexual Psychophysiological Arousal (VESPA)
Acronym: VESPA
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Lori Brotto, Principal Investigator, University of British Columbia
Other Study IDs: H12-01852
Record Dates: First submitted 2012-08-27; First posted 2012-10-04 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Sexual Arousal
Keywords: sexual arousal; pelvic floor sEMG

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: This is an observational study. Women in this study are not receiving any treatments.

SUMMARY:
This study will examine whether measurement of pelvic floor muscle sEMG activity is responsive to explicit sexual stimuli, and whether it correlates with self-reports of sexual arousal in healthy women. Participants' vaginal, labial and anal sEMG readings will be monitored during exposure to neutral, erotic and anxiety-provoking films. Participants will also be required to provide subjective ratings of sexual arousal before and after each film. If pelvic floor sEMG is validated as a psychophysiological measure, these findings may have important clinical and research implications by providing a greater understanding of the mechanisms involved in sexual arousal and for providing a relatively easy method of assessing sexual arousal in a clinical or research setting.

DETAILED DESCRIPTION:
HYPOTHESES:

1. Investigators hypothesize that, relative to the neutral films, PFM EMG activity will significantly increase in response to the erotic film as measured by the labial, anal, and vaginal EMG probes.
2. Investigators hypothesize that, relative to the anxiety-provoking film, PFM EMG activity will significantly increase in response to the erotic film as measured by the labial, anal, and vaginal EMG probes.
3. Investigators hypothesize that continuously measured subjective sexual arousal (via the arousometer) will correlate significantly with PFM EMG activity during the erotic film.

ELIGIBILITY:
Inclusion Criteria:

* Must be female, between the ages of 19-45
* Must be premenopausal
* Must be previously sexually active
* Must be fluent in English

Exclusion Criteria:

* Lack of fluency in English
* Not female between the ages of 19-45
* Not previously sexually active
* Any previous deliveries, either vaginal or by c-section
* Any sexual arousal disorder
* Any genital pain or pelvic pain disorders
* Any bowel or bladder syndromes (e.g. interstitial cystitis, irritable bowel disease, Chron's disease)
* Any urinary incontinence or pelvic organ prolapse
* Undergone medically induced menopause
* Undergone total or partial hysterectomy
* Undergone surgery for incontinence or prolapse
* Using estrogen suppression medication

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy females.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Pelvic floor muscle sEMG activity | This study involves 1 testing session approximately 20 minutes in duration
  Changes in pelvic floor muscle activity in responsive to exposure to explicit sexual stimuli will be assessed using pelvic floor surface electromyography (sEMG).

SECONDARY OUTCOMES:
Sexual Arousal | This study involves 1 testing session approximately 20 minutes in duration
  Self-report sexual arousal will be measured with the Sexual Arousability Inventory (SAI ; Hoon, Hoon, & Wincze, 1976)
Sexual Function | This study involves 1 testing session approximately 20 minutes in duration
  Self-reported sexual function will be measured using the Female Sexual Function Inventory (FSFI; Rosen et al., 2000) and the Derogatis Sexual Functioning Inventory (DSFI; Derogatis & Melisaratos, 1979).

CONTACTS AND LOCATIONS:
Overall Officials: Lori A. Brotto, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Department of Gynaecology, Vancouver, British Columbia, Canada

REFERENCES:
- See also: UBC Sexual Health Lab Website — http://www.obgyn.ubc.ca/SexualHealth/